CLINICAL TRIAL: NCT04666532
Title: Staphylococcus Aureus Translocation From Skin and Nose to Periprosthetic Tissues
Brief Title: S. Aureus Translocation From Skin and Nose to Periprosthetic Tissues
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Rothman Institute Orthopaedics (Other)
Responsible Party: Sponsor
Other Study IDs: JPAR20D165 FARE
Record Dates: First submitted 2020-12-08; First posted 2020-12-14 (Actual); Last update posted 2020-12-14 (Actual); Status verified 2020-12

CONDITIONS: Staphylococcus Aureus
MeSH Terms: conditions — Staphylococcal Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Surgical site infections (SSI) are a significant clinical issue that requires the use of a great amount of resources. In particular, periprosthetic joint infections (PJIs) have potentially catastrophic effects on patients' health-related quality of life, function, healthcare costs, outcomes and medical implications. National surveillance estimates may under-report the true incidence and when considering the large number of total hip (THA) and total knee arthroplasty (TKA) procedures performed each year.

Patients who have a high-level of nasal bacteria have been found to have a risk of surgical site infection that is three to six times the risk compared with noncarriers and low-level carriers. The association between a patient's nasal carriage of S. aureus, specifically MRSA, and PJI has been demonstrated in a systematic review and confirmed in recent cohort studies. While this association seems to be well accepted, no mechanistic explanation has been provided for this association.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing revision total knee or total hip arthroplasty at our institution will be eligible

Exclusion Criteria:

* Patients included in other prospective studies

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants who are undergoing revision total knee or hip arthroplasty by one of the joints surgeons at Rothman Orthopaedics
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2020-10-22 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
S. aureus Culture and Next Generation Sequencing | 1 day
  Diagnostic performance of molecular and culture techniques for S. aureus screening using nasal and groin swabs to determine whether the S. aureus retrieved on the skin and nares of patients who develop a joint infection is identical to the bacteria found in the wound of the PJI

CONTACTS AND LOCATIONS:
Locations (1):
- Rothman Orthopaedic Institute, Philadelphia, Pennsylvania, United States